CLINICAL TRIAL: NCT06708884
Title: Is Telerehabilitation a Good Alternative to Face-to-Face Rehabilitation Beyond Clinical Walls in Recovery After Total Hip Arthroplasty
Brief Title: Telerehabilitation as an Alternative to Face-to-Face Rehabilitation After Total Hip Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Akın Süzer, Principal Investigator, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ErsoyU.22112024
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Total Hip Arthroplasty (THA)
Keywords: total hip arthroplasty; telerehabilitation
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: TR Group (Experimental): TR: telerehabilitation. During the follow-up period, a standard exercise programme will be applied to the TR group via videoconference-based telerehabilitation.
  Interventions: Other: Exercise
- Group 1: F2F Group (Experimental): F2F: face to face. During the follow-up period, a standard exercise programme will be applied to the F2F group via face to face rehabilitation.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — exercise programme will be implemented via telerehabilitation
  Arms: Group 1: TR Group
Other: Exercise — exercise programme will be implemented via face-to-face
  Arms: Group 1: F2F Group

SUMMARY:
The goal of this clinical trial is to learn if telerehabilitation in patients who had undergone total hip arthroplasty. The main questions it aims to answer are:

* Does telerehabilitation improve the functional level of the participants?
* Does telerehabilitation improve the locomotor performance of the participants? Researchers will compare telerehabilitation to face to face rehabilitation (traditional rehabilitation programme) to see if telerehabilitation works in total hip arthroplasty recovery.

Participants will:

* Attend physiotherapy and rehabilitation sessions supervised by a physiotherapist 2 days a week for 8 weeks.
* Participate in assessments (before surgery and at 6 weeks and 12 weeks after surgery).

ELIGIBILITY:
Inclusion Criteria:

* Having hip arthroplasty surgery
* To be able to understand verbal and written information
* No cognitive impairment
* To be able to speak and understand Turkish

Exclusion Criteria:

* Having a neurological disease
* Having a psychiatric disorder
* Visual or hearing loss that cannot be corrected with any assistive device

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Functional level | Assessments will be performed before surgery and at 6 weeks and 12 weeks after surgery.
  Functional level was assessed using the Western Ontario McMaster University Osteoarthritis Index. Western Ontario and McMaster Universities Osteoarthritis Index consists of 24 questions and 3 subcategories (pain, stiffness and physical function). Pain is evaluated with 5 questions, stiffness with 2 questions and physical function with 17 questions. Each question in the Index is scored from 0 (none) to 4 (very severe, very difficult). The total score can be a minimum of 0 and a maximum of 100. In addition, each subcategory can also be evaluated on its own. A higher score on the Index indicates more symptoms and physical disability.

SECONDARY OUTCOMES:
Pain intensity | Assessments will be performed before surgery and at 6 weeks and 12 weeks after surgery.
  Pain intensity was assessed using the pain subcategory of Western Ontario McMaster University Osteoarthritis Index and the Visual Analog Scale. There are 5 questions in the pain subcategory of the Western Ontario and McMaster Universities Osteoarthritis Index. Each question in the Index is scored from 0 (none) to 4 (very severe, very difficult). The pain score can be a minimum of 0 and a maximum of 20. A higher pain score indicates more pain. Visual Analog Scale consists of a horizontal 10 cm straight line. When viewed from left to right, there is a value of 0 at the beginning and 10 at the end of the line. The 0 point of the line indicates no pain and the 10 point indicates the most severe pain felt in life.
Quality of life | Assessments will be performed before surgery and at 6 weeks and 12 weeks after surgery.
  Quality of life will be assessed with the EQ-5D General Quality of Life Questionnaire. The first part of the questionnaire consists of questions related to five different areas of health, including mobility, personal care, usual activities, pain/discomfort, and anxiety/depression. Each question is rated on a three-point scale as 'no problem, some problem and major problem'. Therefore, the questionnaire generates 243 different results. As a result of the scoring, a score between -0.59 and 1 is obtained and 0 indicates death, 1 indicates full health, minus values indicate unconsciousness, etc. The second part of the questionnaire shows the score that the person gives to the health status by marking on a vertical ruler or a thermometer-like visual analogue scale between 0 and 100. A score of 100 indicates the healthiest state.
Locomotor performance | Assessments will be performed before surgery and at 6 weeks and 12 weeks after surgery.
  Locomotor performance was assessed with the stair climb test. Stair Climb Test: The time taken to ascend and then descend a 9-step staircase was recorded as the patient's score.
Lower extremity muscle strength | Assessments will be performed before surgery and at 6 weeks and 12 weeks after surgery.
  Lower extremity muscle strength will be assessed with the a hand dynamometer. Hand Dynamometer: Hip muscles (flexors, extensors, abductors and adductors) and knee extensors will be evaluated using a hand dynamometer (Commander Muscle Tester, JTech, USA). 3 consecutive maximum isometric contraction measurements at 1 minute intervals will be averaged.
Hip Joint Range of Motion (ROM) | Assessments will be performed before surgery and at 6 weeks and 12 weeks after surgery.
  Range of Motion (ROM) will be evaluated by goniometric measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided